CLINICAL TRIAL: NCT02005341
Title: A Prospective, Nonrandomized Study to Assess Lumbar Fusion With Instrumented Posterolateral Gutter Fusions Using NanOss Bioactive
Brief Title: NanOss Bioactive With Autograft and Bone Marrow Aspirate in the Posterolateral Spine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A change in research priorities after a merger
Sponsor: Pioneer Surgical Technology, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 2010-02b
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Lumbar Spinal Stenosis Secondary to Other Disease
Keywords: Lumbar; fusion
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autograft bone (Active Comparator)
  Interventions: Device: Autograft
- nanOss with bone marrow aspirate (Experimental)
  Interventions: Device: nanOSS

INTERVENTIONS:
Device: nanOSS
  Arms: nanOss with bone marrow aspirate
Device: Autograft
  Arms: Autograft bone

SUMMARY:
The purpose of this study is to assess lumbar fusion using nanOss Bioactive bone void filler

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 21 years of age and skeletally mature.
2. Must have cervical disc disease (defined as neck pain of discogenic origin with degeneration of the disc confirmed by history and radiographic studies) at one level in the cervical spine between C3 to T1.
3. Must have completed a minimum of six weeks of unsuccessful conservative, non-operative care or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of conservative treatment.
4. Has pre-operative objective evidence of primary diagnosis confirmed by appropriate imaging studies (Anteroposterior/Lateral/Flexion/Extension X-rays & a recent MRI).
5. Is willing and able to comply with all clinical investigation visits and procedures including screening treatment procedures, post-operative management, the follow-up schedule and completion of forms or questionnaires.
6. Is able to understand and sign the patient information sheet/informed consent form.

Exclusion Criteria:

1. Requires fusion at more than one level.
2. Has had prior fusion at the level to be treated.
3. Has a metabolic or systemic bone disorder.
4. Has a disease that significantly inhibits bone healing (i.e., severe osteoporosis, osteomalacia, Paget's disease).
5. Has a systemic or local infection (active or latent).
6. Has acute or chronic infections in the surgical area (i.e., soft tissue infections; inflammatory, bacterial bone disorders, osteomyelitis).
7. Chronic use of steroids, other than episodic use or inhaled corticosteroids.
8. Has any significant general illness (i.e., HIV, active metastatic cancer of any type, uncontrolled diabetes Type I, dialysis dependent renal failure, symptomatic liver disease).
9. Has a mental or physical condition that would limit the ability to comply with study requirements or would preclude accurate evaluation.
10. Is immunocompromised or being treated with immunosuppressive agents (including chemotherapy or radiation treatment).
11. Has documented allergies to hydroxyapatite or porcine collagen, PEEK, titanium, titanium alloy or tantalum.
12. Is currently pregnant, or interested in becoming pregnant during the clinical investigation follow-up.
13. Is a smoker.
14. Is non-English speaking.
15. Requires the use of a bone-growth stimulator.
16. Is a prisoner.
17. Is currently involved in another drug or device clinical investigation that may confound the clinical trial investigation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Fusion at 12 months postoperatively. | 12 months

IPD SHARING:
Plan to Share IPD: No